CLINICAL TRIAL: NCT00496158
Title: A Multi-Center, Randomized, Double-Blind, Active-Control, 96 Week, Phase III Trial of the Efficacy and Safety of Clevudine Compared With Adefovir at Weeks 48 and 96 in Nucleoside Treatment-Naïve Patients With HBeAg Negative Chronic Hepatitis Due to Hepatitis B Virus
Brief Title: Efficacy and Safety of Clevudine Compared With Adefovir in Patients With Chronic Hepatitis Due to Hepatitis B Virus
Acronym: QUASH2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated in the interest of patient safety.
Sponsor: Pharmasset (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CI-PSI-5268-06-306
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Chronic Hepatitis; Hepatitis B
Keywords: Nucleoside Treatment-Naïve Patients with HBeAg Negative Chronic Hepatitis due to Hepatitis B Virus; hepatitis b virus
MeSH Terms: conditions — Hepatitis, Chronic; Hepatitis B | interventions — clevudine; adefovir

INTERVENTIONS:
Drug: Clevudine
Drug: Adefovir

SUMMARY:
The objectives of this study are to compare in nucleoside treatment-naïve subjects, the efficacy and safety of clevudine 30 mg once daily versus adefovir 10 mg once daily, each as monotherapy, for 48 weeks, 72 weeks, and 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Nucleoside treatment-naïve subjects of either gender, females who are non-pregnant and non-lactating, aged 16 years or older (or the legal age of consent as allowed by local regulations), with compensated hepatic function despite a diagnosis of chronic HBeAg negative hepatitis B infection (i.e., based on serological, virological and histological markers) will be eligible for this study.
* Subjects entering the study with an historical biopsy will have chronic hepatic inflammatory injury at screening (Knodell HAI score ≥ 4 and modified Ishak fibrosis score ≤ 5).
* The number of subjects entering the study with an Ishak fibrosis score of 5 will be limited to approximately 10%. If applicable, subjects must cease previous treatment with any form of alpha interferon 12 months prior to baseline.
* For eligibility, subjects must meet the laboratory criteria for total bilirubin, prothrombin time, serum albumin, platelet count, absolute neutrophil count, ANA titer and have a creatinine clearance of ≥ 50 mL/min.

Exclusion Criteria:

* Subjects participating in a clinical trial or receiving an investigational agent for any reason within 60 days of baseline will be excluded.
* Subjects with clinically significant concomitant diseases will be excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-08

CONTACTS AND LOCATIONS:
Overall Officials: M Michelle Berrey, MD, MPH, Study Director — Pharmasset
Locations (115):
- United States (59):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Anaheim, California
  - Advanced Clinical Research Institution, Anaheim, California
  - Fresno, California
  - West Gastroenterology Medical Group, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Los Angeles, California
  - San Clemente, California
  - Sharp Rees-Stealy Medical Group, Inc., San Diego, California
  - Medical Associates Research Group, San Diego, California
  - San Diego, California
  - San Francisco, California
  - California Pacific Medical Center, San Francisco, California
  - Quest Clinical Research, San Francisco, California
  - Ucsf/Sfgh, San Francisco, California
  - San Mateo Medical Center, San Mateo, California
  - The William W. Backus Hospital, Norwich, Connecticut
  - North Miami Beach, Florida
  - Tampa, Florida
  - Infectious Disease Reseach Institute, Inc, Tampa, Florida
  - Liver Center, Honolulu, Hawaii
  - Iowa Health-Des Moines, Des Moines, Iowa
  - Tulane Medical Center, New Orleans, Louisiana
  - New Orleans, Louisiana
  - Banks Hepatology Institute, College Park, Maryland
  - Boston, Massachusetts
  - Digestive Health Specialists, Tupelo, Mississippi
  - Saint Louis University, St Louis, Missouri
  - Hillsborough, New Jersey
  - UMA Research Department, Binghamton, New York
  - Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - VAMC/NYU, New York, New York
  - Weill Cornell Medical College, New York, New York
  - New York, New York
  - Asheville, North Carolina
  - Asheville Gastroenterology, Asheville, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Portland, Oregon
  - The Oregon Clinic P.C., Portland, Oregon
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Nashville Gastrointestinal Specialists, Inc, Nashville, Tennessee
  - Austin, Texas
  - Austin Gastroenterology, PA, Austin, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Methodist Transplant Physicians, Dallas, Texas
  - Galveston, Texas
  - Advanced Liver Therapies, Houston, Texas
  - Century Clinical Research Inc, Houston, Texas
  - Brooke Army Mecial Center, San Antonio, Texas
  - Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Fairfax, Virginia
  - Metropolitan Research, Fairfax, Virginia
  - Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Tacoma, Washington
- Argentina (10):
  - Centro de Hepatologia, Buenos Aires
  - Funcei, Buenos Aires
  - Fundacion Favaloro, Buenos Aires
  - Hospital Aleman, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Hospital Universitario Austral, Buenos Aires
  - Sanatorio de la Trinidad Mitre, Buenos Aires
  - Sanatorio Guemes, Buenos Aires
  - Sanatorio Dei Salvador, Córdoba
  - H.I.G.A O. Alende, Mar del Plata
- Australia (10):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St. Vincent's, Fitzroy, Victoria
  - Western Hospital, Footscray, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Canada (9):
  - University of Calgary, Calgary, Alberta
  - Liver and Intestinal Research Center (LAIR Center), Vancouver, British Columbia
  - UBC/ Downtown ID Clinic, Vancouver, British Columbia
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
- China (3):
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - The Chinese University of Hong Kong, Hong Kong
  - The University of Hong Kong, Hong Kong
- Greece (3):
  - Agios Savvas Hospital, Athens
  - Ippokration General Hospital, Athens
  - Laiko General Hospital, Athens
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico
- Spain (7):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
- Taiwan (5):
  - Chang Gung Memorial Hospital Kaosiung, Kaohsiung City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
- Thailand (6):
  - NKC Institute of Gastroenterology and Hepatology/ Songklanagarind Hospital, Hat Yai, Changwat Songkhla
  - Phramongkutklao Hospital, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok
  - Chiang Mai University, Chiang Mai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
  - Naresuan University, Phitsanulok
- United Kingdom (2):
  - Gartnavel General Hospital, Glasgow
  - St. George's NHS Trust, London